CLINICAL TRIAL: NCT01319617
Title: Evaluation of SENSIMED Triggerfish Safety and Tolerability in Glaucoma Patients and Glaucoma Suspects
Brief Title: SENSIMED Triggerfish Safety and Tolerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/05
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish (Experimental)
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Soft contact lens-based device intended for continuous recording of relative changes in IOP

SUMMARY:
The purpose of this investigation is to study the safety and tolerability of SENSIMED Triggerfish, a soft contact lens-based device intended to continuously record relative changes in intraocular pressure (IOP). The investigation enrols glaucoma patients and glaucoma suspects. All subjects receive two 24-hour recording sessions with the device in an ambulatory setting and at weekly interval. The level of discomfort in the study eye after 24 hours and side effects are the main endpoints of the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comply with the study procedures
* Subject is 18-80 years old
* Glaucoma patient, with glaucomatous optic neuropathy based on clinical assessment of stereoscopic optic disc photographs and/or repeatable abnormal standard automated perimetry (SAP) visual fields at baseline, defined as a pattern standard deviation with P<0.05 or a glaucoma Hemifield test "outside normal limits
* Glaucoma suspect, with suspicious optic disc appearance (as determined by subjective assessment on the baseline visit) or elevated IOP (>21 mmHg) but normal and reliable SAP visual fields at baseline
* Subject has consented to be in the trial and signed informed consent is available before any study related procedures are carried out
* Visual acuity of 20/200 or better in the study eye
* Ability of subject to understand the character and individual consequences of the study
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Subjects with contraindications for wearing contact lenses
* Severe dry eye syndrome
* Keratoconus or other corneal abnormality
* Conjunctival or intraocular inflammation
* Eye surgery prior to and throughout the study, except prior uncomplicated cataract surgery a minimum of 3 months prior to the investigation
* Full frame metal glasses during SENSIMED Triggerfish® recording
* Known hypersensitivity to silicone, plaster or ocular anesthesia
* Pregnancy and lactation
* Simultaneous participation in other clinical studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Medeiros, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Mansouri K, Medeiros FA, Tafreshi A, Weinreb RN. Continuous 24-hour monitoring of intraocular pressure patterns with a contact lens sensor: safety, tolerability, and reproducibility in patients with glaucoma. Arch Ophthalmol. 2012 Dec;130(12):1534-9. doi: 10.1001/jamaophthalmol.2013.1350. PMID 23229696
- [Derived] Mansouri K, Liu JH, Weinreb RN, Tafreshi A, Medeiros FA. Analysis of continuous 24-hour intraocular pressure patterns in glaucoma. Invest Ophthalmol Vis Sci. 2012 Dec 13;53(13):8050-6. doi: 10.1167/iovs.12-10569. PMID 23139273
- [Derived] Mansouri K, Medeiros FA, Tafreshi A, Weinreb RN. Continuous 24-hour monitoring of intraocular pressure patterns with a contact lens sensor: safety, tolerability, and reproducibility in patients with glaucoma. Arch Ophthalmol. 2012 Dec;130(12):1534-9. doi: 10.1001/archophthalmol.2012.2280. PMID 22892888

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from medical clinic from January to September 2011
Groups:
- SENSIMED Triggerfish: SENSIMED Triggerfish is a device containing a soft silicone contact lens sensor detecting ocular dimensional changes related to IOP through an integrated strain gauge. The device energy and data transfer between the contact lens sensor and the external recording and data storage unit is done using telemetry.
  All study subjects received SENSIMED Triggerfish on one eye for 24 hours at two occasions in ambulatory mode, without restriction of activities apart from those contraindicated by the device instructions for use. The device was installed and removed by the study staff during visits to the study center.
Period: Overall Study
Arm/Group | SENSIMED Triggerfish
Started | 41
Completed | 40
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 54.6 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Ocular Discomfort
Description: Ocular discomfort in the study eye is reported by patients on a 100-mm visual analog scale (left end 0 mm, no discomfort; right end 100 mm, very severe discomfort) as the distance from the left end to the patient's mark after wearing the device for 24 hours at two occasions separated by one week. Values for both sessions were averaged.
Time Frame: After 24 hours of device wear
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 40
mm | 25.5 (18.6)

ADVERSE EVENTS:
Arm/Group | SENSIMED Triggerfish
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 39/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SENSIMED Triggerfish (N=41)
conjunctival edema (Eye disorders) | 1 (1)
device intolerance (Eye disorders) | 1 (1)
eye irritation (Eye disorders) | 3 (3)
eye pressure mark (Eye disorders) | 13 (17)
eye pruritus (Eye disorders) | 3 (3)
ocular discomfort (Eye disorders) | 1 (2)
ocular hyperemia (Eye disorders) | 32 (56)
punctate keratitis (Eye disorders) | 6 (6)
vision blurred (Eye disorders) | 33 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No